CLINICAL TRIAL: NCT06106490
Title: Addition of Pulsed Radiofrequency to Suprascapular Nerve Block With Glenohumeral Steroid Injection in Patients With Chronic Shoulder Pain
Brief Title: Pain Managment in Chronic Shoulder Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nahla yahia, assistant lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FMASU MD128/2023
Record Dates: First submitted 2023-10-14; First posted 2023-10-30 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Pain Management
Keywords: Shoulder pain; Suprascapular nerve block; Pulsed radiofrequency
MeSH Terms: conditions — Shoulder Pain | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suprasacapular nerve block (Active Comparator): Patients will receive ultrasound guided intra articular Gleno-humeral steroid injection of Diprofos® (betamethasone 14 mg/ 2ml) and ultrasound guided suprascapular nerve block US SSN with 10mL of 0.25% preservative-free bupivacaine
  Interventions: Other: the effect of adding pulsed radiofrequency (PRF) modality to suprascapular nerve injection with ultrasound glenohumeral steroid in chronic shoulder pain patients
- Pulsed Radiofrequency group (Active Comparator): Patients will receive ultrasound guided intra articular Gleno-humeral steroid injection of Diprofos® (betamethasone 14 mg/ 2ml) and ultrasound guided suprascapular nerve block US SSN with 10mL of 0.25% preservative-free bupivacaine with application of pulse PRF at 42 Celsius of suprascapular nerve for 480 seconds.
  Interventions: Other: the effect of adding pulsed radiofrequency (PRF) modality to suprascapular nerve injection with ultrasound glenohumeral steroid in chronic shoulder pain patients

INTERVENTIONS:
Other: the effect of adding pulsed radiofrequency (PRF) modality to suprascapular nerve injection with ultrasound glenohumeral steroid in chronic shoulder pain patients — Suprascapular nerve block group: Patients will receive ultrasound guided intra articular Gleno-humeral steroid injection of Diprofos® (betamethasone 14 mg/ 2ml) and ultrasound guided suprascapular nerve block US SSN with 10mL of 0.25% preservative-free bupivacaine
  Pulsed radiofrequency group: Patients will receive ultrasound guided intra articular Gleno-humeral steroid injection of Diprofos® (betamethasone 14 mg/ 2ml) and ultrasound guided suprascapular nerve block US SSN with 10mL of 0.25% preservative-free bupivacaine with application of pulse PRF at 42 Celsius of suprascapular nerve for 480 seconds.

SUMMARY:
The purpose of this study is to evaluate the effect of adding pulsed radiofrequency (PRF) modality to suprascapular nerve injection with ultrasound glenohumeral steroid in chronic shoulder pain patients focusing on both changes in pain and function scores

DETAILED DESCRIPTION:
Shoulder pain is the second most prevalent musculoskeletal condition in adults which is frequently treated poorly and results in chronic pain .

The use of steroid injection has been demonstrated to be superior to conventional therapies, particularly non-steroidal anti-inflammatory drugs. Its impact is transient (4-6 weeks) and occasionally may not be clinically sufficient .

An alternate analgesic injection for the pain management of numerous shoulder diseases is the suprascapular nerve block (SSN) .

Although pulse radiofrequency analgesia typically lasts for a much longer period than nerve blocking, it has become increasingly popular to apply pulse radiofrequency to peripheral nerves.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged from 21-60 years.
* Patients with American Society of Anesthesiologists (ASA) physical status I and II.
* Chronic shoulder pain (>3 months) and will undergo interventional treatment due to inadequate response to conservative treatments.

Exclusion Criteria:

* Refusal of procedure or participation in the study by patients.
* History of shoulder surgery, another intervention history between 3 months before and 1 year after the intervention applied.
* Patients with chronic pain syndrome due to other shoulder pathology (fibromyalgia, cervical discopathy, brachial plexus injury).
* Uncontrolled diabetes mellitus patients with glycated hemoglobin (HbA1C) levels of more than 7%.
* Patients with known history of allergy to the study drugs.
* Infection at site of injection.
* Cognitive or psychiatric illness that will lead to inability to cooperate, speak, or provide informed consent.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
change of Shoulder Pain and Disability Index (SPADI) questionnaire in both groups after the intervention | 15th day, 1st month, 3rd month and 6th month
  The Shoulder Pain and Disability Index (SPADI) a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities, overall total scores range from 0 to 130 with a percentage score of 0 indicating less shoulder disability and 100 indicating more shoulder dysfunction

SECONDARY OUTCOMES:
Numerical pain rating scale (NRS).physiological parameter | 15th day, 1st month, 3rd month and 6th month
  patients are asked to circle the number between 0 and 10, 0 and 20 or 0 and 100 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Duration of pain relief physiological parameter | 15th day, 1st month, 3rd month and 6th month
  when the effect of the intervention will be lost after the intervention
Active range of motion (AROM).physiological parameter | 15th day, 1st month, 3rd month and 6th month
  will be measured using a geniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Amr Abdelfatah, proffessor, Study Director — Ainshams University
Locations (1):
- Faculty of medicine Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
summary results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: one year after publication
Access Criteria: internet search by keywords